CLINICAL TRIAL: NCT00002689
Title: Phase II Interstitial Colloidal 32P Integrated in The Treatment of Non-Resectable Pancreatic Cancer
Brief Title: Radiation Therapy Plus Chemotherapy in Treating Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for Molecular Medicine (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CMM-95079; CDR0000064415 (Registry Identifier: PDQ (Physician Data Query)); CH/UMC-95079; NCI-V95-0760
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2007-06

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Dexamethasone; Fluorouracil; Brachytherapy; Phosphorus-32; Radiotherapy

INTERVENTIONS:
Drug: dexamethasone
Drug: fluorouracil
Radiation: brachytherapy
Radiation: phosphorus P32
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy combined with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of brachytherapy followed by external-beam radiation therapy plus chemotherapy in treating patients who have pancreatic cancer that cannot be removed surgically.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response/remission rate, survival, and degree of local control from interstitial colloidal phosphorus P32 followed by external beam radiotherapy and chemotherapy in patients with unresectable pancreatic cancer.

OUTLINE: Patients are stratified according to prior therapy (yes vs no).

Patients receive dexamethasone intratumorally, then macroaggregated albumin and interstitial phosphorus P32 intratumorally. Most patients receive a second course of this brachytherapy.

Patients then proceed to chemoradiotherapy beginning 7-14 days after brachytherapy. Radiotherapy is administered 5 days a week for 6.4 weeks. Fluorouracil IV is administered every other day for 4 doses during weeks 1 and 2.

Patients are followed monthly for 1 year then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven unresectable adenocarcinoma of the pancreas limited to the head, body, or tail of the pancreas

  * Diameter no greater than 5 cm
  * Volume no greater than 66 mL
* No ascites (with or without tumor cells)
* No endoscopically proven tumor penetration of duodenum or stomach

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Hematopoietic:

* WBC at least 3,000/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9 g/dL (transfusion allowed)

Hepatic:

* No hepatic disease
* At least 50% uptake of technetium-sulfur colloid in normal liver if cirrhosis suspected
* No vascular occlusion of portal system

Renal:

* Creatinine no greater than 1.5 mg/dL
* BUN no greater than 25 mg/dL

Other:

* No Crohn's disease, ulcerative colitis, or other inflammatory bowel disease
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* If prior chemotherapy, test dose of colloidal phosphorous P32 administered prior to attempted treatment

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to pancreas, liver, or upper gastrointestinal tract

Surgery:

* No complete surgical resection
* No splenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 1995-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Response rate
Duration of remission
Survival

SECONDARY OUTCOMES:
Patterns of failure

CONTACTS AND LOCATIONS:
Overall Officials: Stanley E. Order, MD, ScD, FACR, Study Chair — Center for Molecular Medicine
Locations (2):
- United States (2):
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Center for Molecular Medicine, Garden City, New York